CLINICAL TRIAL: NCT03320122
Title: School-Based Tele-Physiatry Assistance for Rehabilitative and Therapeutic Services for Children With Special Health Care Needs Living in Rural and Underserved Communities
Brief Title: School-Based Tele-Physiatry Assistance for Rehabilitative and Therapeutic Services
Acronym: STARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 994055
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Pediatrics; Physical and Rehabilitation Medicine; Physical Therapy Modalities
Keywords: Telemedicine
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: The proposed program will target MTUs and patients in counties were pediatric physiatrists and other multidisciplinary team members are underrepresented. In this proposed model, the investigators will randomly select at least 350 patient encounters: approximately 175 children will receive care using tele-physiatrist medical direction; 101 children will receive care from a pediatric physiatrist who travels to the MTU to provide in-person care; and 74 children will receive care under a non-pediatric specialist's medical directorship. Once the care model has been created at each site, patients from each cohort will be selected using a clustered, clinic based randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telemedicine (Experimental): Medical Direction will be provided by pediatric physiatrists using telemedicine.
  Interventions: Other: Telemedicine
- In-Person Pediatric Physiatrist (Active Comparator): Medical Direction will be provided by pediatric physiatrists in-person.
  Interventions: Other: In-Person Pediatric Physiatrist
- In-Person Non-Pediatric Physiatrist (Active Comparator): Medical Direction will be provided by contracted physicians (i.e., non-pediatric physiatrists) in-person care.
  Interventions: Other: In-Person Non-Pediatric Physiatrist

INTERVENTIONS:
Other: Telemedicine — Medical direction will be provided to MTUs through a video-based conferencing unit. Each telemedicine unit includes a Rubbermaid medical grade cart with a Polycom RealPresence 500 Series high-resolution video-conferencing unit flat screen to display video. Each cart also comes with an Uninterrupted Power Supply (UPS) to make the unit mobile if needed or to properly shut it down in the event of power failure.
  Arms: Telemedicine
Other: In-Person Pediatric Physiatrist — UC Davis pediatric physiatrists will drive out to the school-based MTUs to provide medical direction in person.
  Arms: In-Person Pediatric Physiatrist
Other: In-Person Non-Pediatric Physiatrist — A contracted physician (i.e., a non pediatric physiatrist) would provide medical direction in person.
  Arms: In-Person Non-Pediatric Physiatrist

SUMMARY:
Using a randomized trial design, the goal of this project is to prospectively compare outcomes from a telemedicine-based model of care to two cohorts: patients who receive in-person pediatric physiatrist medical direction (the "gold standard"), and those who receive medical oversight from non-specialist community providers. This project will determine the impact of this new model of care using telemedicine on parent/guardian satisfaction, adherence rates to an evidence-based hip surveillance program, and economic efficiency.

DETAILED DESCRIPTION:
During this study, a novel model of care will be developed and tested using telehealth technologies to bring necessary medical expertise to children with special health care needs living in rural and underserved communities. This model of care will be implemented in eight school-based Medical Therapy Units (MTUs) in northern California using a randomized design. The investigators hypothesize that this model of care will result in 1) equal satisfaction of the care received in-person from pediatric physiatrists and increased satisfaction of the care received from non-pediatric specialists; 2) equal adherence rates to an evidence-based hip surveillance program when compared to children who receive care from in-person pediatric physiatry care and better adherence than children who receive care from non-pediatric specialists; and 3) cost savings when compared to medical direction provided in-person by pediatric physiatrists and non-pediatric specialist providers.

The first 6 months of the project will be a "ramp-up" period during which the protocol will be re-reviewed during MTU site visits and necessary contracts and approvals will be in place. The last 6 months will be reserved for data analysis, study closeout, and manuscript preparation. The intervention phase will include various designs of implementation. For those schools currently without pediatric physiatry services, the investigators will provide MTU services using telemedicine and add in-person clinics. For those schools where medical direction is provided by non-pediatric physiatrists, the investigators will augment current services using telemedicine to provide medical direction to some children using pediatric physiatrists. For those schools where pediatric physiatrists travel long distances to provide medical direction during scheduled clinics, the investigators will similarly add additional telemedicine services such that an augmented mixed model of in-person and telemedicine pediatric physiatrist medical direction will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include children with special health care needs enrolled in the CCS Medical Therapy Program receiving care at one of the participating sites during the study period.

Exclusion Criteria:

* Children with special health care needs not enrolled in the CCS Medical Therapy Program.

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 350 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Parent/Guardian Satisfaction Survey | Over 1 day for each patient
  The effect of providing pediatric physiatrist medical direction across groups will be measured through satisfaction surveys that will be distributed to participating parents and guardians. Satisfaction surveys will utilize a seven-point Likert scale and the investigators will assess the inter-item reliability, dimensionality and construct validity of satisfaction scales using standard multivariable analysis techniques. A higher score represents a higher satisfaction rate. The investigators postulate that a minimally important clinically significant difference is approximately 0.50 points, while a difference of 0.30 is tolerably close for purposes of non-inferiority.
Evidence-Based Hip Surveillance Program Survey | Over 1 day for each patient
  The hip surveillance survey utilizes several Yes/No responses to compare guideline adherence between the three cohorts and the questions are directly linked to the clinical expectations and explicit guidelines for the appropriate timing and frequency of x-rays and exams. Adherence rates will be compared by adjusted odds ratios.
European Quality of Life-5 Dimensions (EQ-5D) Survey | Over 1 day for each patient
  The EQ-5D is a quality of life assessment tool for measuring "utility." The "utility" is a comprehensive health measure, ranging from 0 (death) to 1 (perfect health), based on an individual's health state in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The utility for a certain health condition is calculated by applying an established formula that assigns weights to each of the levels in each dimension determined by this health condition. These data on a quality of life will be used in a cost-effectiveness analysis.
Economic Efficiency | Up to 4 years
  Cost analysis will estimate cost changes resulting from the introduction of this new model of care from the perspectives of patients and families, physicians and healthcare providers, and payers. The proposed economic evaluative methods will integrate all of the effectiveness results from patient encounter data and EQ-5D survey data. Cost analysis will estimate return-on-investment indicating the cost-saving amount per $1 investment in telemedicine compared to MTUs without telemedicine.

CONTACTS AND LOCATIONS:
Overall Officials: James Marcin, MD, MPH, Principal Investigator — UC Davis Health
Locations (1):
- University of California, Davis, Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-satisfaction-with-school-based-telemedicine-574952/